CLINICAL TRIAL: NCT06234839
Title: Efficacy of Two Orally Administered Lactobacillus Reuteri Strains for Gingivitis Reduction in Young Adults: A Randomized Controlled Clinical Trial
Brief Title: Lactobacillus Reuteri Strains for Gingivitis Reduction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Autonoma de San Luis Potosí (Other)
Responsible Party: Principal Investigator, José Arturo Garrocho Rangel, Proffesor/Lecturer/Reasearcher, Universidad Autonoma de San Luis Potosí
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LLeuteri220124
Record Dates: First submitted 2024-01-22; First posted 2024-01-31 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Gingival Inflammation
Keywords: Gingivitis; Lactobacillus reuteri; Bacteriotherapy; Clinical randomized trial
MeSH Terms: conditions — Gingivitis

STUDY DESIGN:
Intervention Model Description: Both study groups underwent conventional mechanical periodontal therapy/oral anti-plaque hygiene. However, the experimental group additionally received the administration of two daily tablets, containing both L. reuteri strains, for 30 days, while the control group did not.
Who Masked: Outcomes Assessor
Masking Description: The clinical evaluators of the results were unaware that each patient belonged to one of the 2 study groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Probiotic group (Experimental): The experimental group received conventional mechanical periodontal therapy and oral anti-plaque hygiene training, plus the administration of two daily tablets, containing both L. reuteri strains, for 30 days.
  Interventions: Dietary Supplement: L. reuteri (DSM 17938 and ATCC PTA 5289) in form of oral tablets
- No probiotic group (No Intervention): The control group also received conventional mechanical periodontal therapy and oral anti-plaque hygiene training; however, this group did not receive the administration of the probiotic tablets.

INTERVENTIONS:
Dietary Supplement: L. reuteri (DSM 17938 and ATCC PTA 5289) in form of oral tablets — Each subject of the experimental group was instructed to dissolve inside the mouth two tablets per day (in the morning and before going to bed at night), during the experimental period of 30 days. The tablets were provided by BioGaia ProDentis® (Stockholm, Sweden). The tablets contained two strains of L. reuteri (DSM-17938 and ATCC PTA 5289), at a dose of 2 x 108 CFU/tablet.
  Other Names: Conventional mechanical periodontal therapy and oral anti-plaque hygiene training
  Arms: Probiotic group

SUMMARY:
The aim of the present study was to investigate the potential beneficial effects in volunteer young adults of orally administered L. reuteri (DSM 17938 and ATCC PTA 5289) on gingival inflammation. The null hypothesis was that no difference would be manifested by probiotic therapy regarding the conventional mechanical treatment (without probiotic administration).

DETAILED DESCRIPTION:
Aim. To investigate the potential beneficial effects in volunteer young adults of orally daily administered L. reuteri (DSM 17938 and ATCC PTA 5289) on gingival inflammation. The null hypothesis was that no difference would be manifested by probiotic therapy regarding the conventional mechanical treatment (without probiotic administration).

Methods. A randomized controlled parallel clinical trial was conducted in sixty young adults (18-35 yrs old) with chronic marginal gingivitis for one month. Initially, both study groups underwent conventional mechanical periodontal therapy/oral anti-plaque hygiene. However, the experimental group additionally received the administration of two daily tablets, containing both L. reuteri strains, for 30 days, while the control group did not. Different clinical outcome variables (plaque (PI) and gingival (GI) indices, bleeding on probing (BOP), and crevicular fluid volume (CFV)) were recorded and compared between the study groups, both at baseline and at the end of the interventions, 30 days later. Statistical descriptive and inferential tests were performed (data distribution normality, Student's t, and Wilcoxon-Mann-Whitney tests).

ELIGIBILITY:
Inclusion Criteria:

* Non-smokers (at least for the last 6 months).
* Initial mean gingival index (GI) between 1.5 - 2.
* With a minimum of 20 teeth present in the oral cavity.

Exclusion Criteria:

* Periodontal pockets > 4 mm.
* Recent intake of antibiotics or anti-inflammatory drugs and/or reception of dental prophylaxis.
* Daily consumption of analgesics, probiotics, or oral antimicrobial rinses/gels.
* Overweight (MCI >25).
* Alcohol or recreative drug frequent consumers.
* Pregnancy or breast-feeding.
* Allergy or hypersensitivity to study products
* Fixed orthodontic appliances.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2023-01-07 (Actual); Primary Completion 2023-07-18 (Actual); Study Completion 2023-12-06 (Actual)

PRIMARY OUTCOMES:
Gingival index | 0, 7, 14, 21 and 30 days.
  The Gingival Index (GI) scores each site on a 0 to 3 scale, with 0 being normal and 3, being severe inflammation characterized by edema, redness, swelling, and spontaneous bleeding.
Plaque index | 0, 7, 14, 21 and 30 days.
  The plaque index assesses the amount of dental plaque visible on the vestibular and lingual surfaces of all teeth, except the third molars. The bacterial plaque developer solution was used to define cumulative amounts of plaque with criteria from 0 to 5.
Bleeding on probing | 0, 7, 14, 21 and 30 days.
  BOP describes bleeding induced by gentle manipulation of the tissue. The probing is typically completed to the depth of the gingival sulcus, or the area between the gingiva and the tooth.
Crevicular fluid volume | 0, 7, 14, 21 and 30 days.
  Gingival crevicular fluid is an inflammatory exudate derived from the periodontal tissues. It is composed of serum and locally generated materials such as tissue breakdown products, inflammatory mediators, and antibodies directed against dental plaque bacteria.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Universidad Autónoma de san Luis Potosi, San Luis Potosí City, Mexico

IPD SHARING:
Plan to Share IPD: No